CLINICAL TRIAL: NCT02708966
Title: Effect of the Administration of Gymnema Sylvestre on Glycemic Control, Insulin Secretion and Insulin Sensitivity in Patients With Impaired Glucose Tolerance.
Brief Title: Effect of Gymnema Sylvestre on Patients With Impaired Glucose Tolerance.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Esperanza Martínez-Abundis, PHD, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GSIG
Record Dates: First submitted 2016-03-10; First posted 2016-03-15 (Estimated); Results first posted 2020-11-18 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Impaired Glucose Tolerance
Keywords: Gymnema Sylvestre; Glycemic control
MeSH Terms: conditions — Glucose Intolerance | interventions — Gurmarin protein, Gymnema sylvestre

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gymnema Sylvestre (Experimental): Patients with IGT
  Interventions: Drug: Gymnema Sylvestre
- Placebo (Placebo Comparator): Patients with IGT
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gymnema Sylvestre — Gymnema Sylvestre, 300mg capsules 2 times daily with the first bite of breakfast and dinner
  Other Names: Gurmar
  Arms: Gymnema Sylvestre
Drug: Placebo — Placebo, 300mg capsules 2 times daily with the first bite of breakfast and dinner
  Other Names: Calcined Magnesia
  Arms: Placebo

SUMMARY:
Prediabetes (PD) was defined as an state in which glucose levels are above normal but not enough to meet criteria for the diagnosis of type 2 diabetes (T2D). PD can be presented as impaired fasting glucose (IFG), impaired glucose tolerance (IGT) and glycated hemoglobin A1c (A1C) altered. The International Diabetes Federation (IDF) reported that in 2013 the prevalence of IGT was 6.9% which is equivalent to approximately 316 million individuals with IGT, it is expected that by 2035 this number will increase to 417 million people affected. Many hypoglycemic effects attributed to Gymnema sylvestre have been reported, including: increase of insulin secretion, regeneration of pancreatic islet cells, increased glucose utilization in various ways and inhibition of glucose uptake in the intestine.

DETAILED DESCRIPTION:
The target is to evaluate the effect of the administration of Gymnema Sylvestre on glycemic control, insulin secretion and insulin sensibility on patients with IGT. The investigators will conduct a double-blind trial, randomized, placebo control group, each group 12 female and male patients, between 30 and 59 years old with IGT (2-h values in the oral glucose tolerance test, OGTT) from 140 mg / dL to 199 mg / dL), Body Mass Index (BMI) from 25 to 34.9 kg / m2. Randomization will determine who will receive the intervention during the 9-week trial (Gymnema Sylvestre capsules, 300 mg 2 times daily with the first bite of breakfast and dinner or homologated placebo capsules). The clinical findings and laboratory tests include a metabolic profile and biosafety, which will be made at baseline and at week 9. Body weight, body fat, BMI and blood pressure will be determined during the initial and final visit. Adverse events and adherence to treatment will be documented. Statistical analysis: Mann-Whitney U test, Wilcoxon and Fisher exact test. It is considered with significance at p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 25.0-34.99 kg / m2.
* Diagnosis of IGT (2h-OGTT Values between 140mg / dl and 199mg / dl.)
* Written informed consent.
* body weight stable over the last 3 months.
* Women in follicular phase of the menstrual cycle (days 3 to 8 of the cycle) at the time of laboratory tests.
* Women who are not contemplated get pregnant within the next 6 months.

Exclusion Criteria:

* Women pregnant or breastfeeding.
* Physical or mental disability that makes it impossible to perform the intervention.
* Diagnosis of hypertension or heart failure.
* Smokers.
* Untreated thyroid disease.
* Consumption of oral agents or other medications or supplements with proven properties that modify the behavior of glucose and lipids (oral hypoglycemic agents, insulin, lipid-lowering).
* Diagnosis of liver disease or elevation twice of the upper normal value of liver enzymes.
* Diagnosis of renal disease or creatinine > 1.5 mg / dl.
* Diagnosis of Type 2 Diabetes Mellitus (T2DM) Fasting glucose ≥ 126 mg / dL and/or 2h-OGTT ≥ 200 mg / dL and/or A1C ≥ 6.5%.
* Total Cholesterol ≥ 280 mg/dL.
* Triglycerides ≥ 300 mg/dL.
* Known allergy to calcined magnesia or Gymnema sylvestre.

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03; Primary Completion 2018-09 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esperanza Martínez-Abundis, PhD, Principal Investigator — Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara
Locations (1):
- Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara, Guadalajara, Jalisco, Mexico

RESULTS

PARTICIPANT FLOW:
Groups:
- Gymnema Sylvestre: Patients with impaired glucose tolerance (IGT)
  Gymnema Sylvestre: Gymnema Sylvestre, 300mg capsules 2 times daily with the first bite of breakfast and dinner
Period: Overall Study
Arm/Group | Gymnema Sylvestre | Placebo
Started | 15 | 15
Completed | 13 | 13
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gymnema Sylvestre | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47 (10) | 44 (7) | 45 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 15 | 30
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 15 | 15 | 30
Body Weight (BW) [Mean (Standard Deviation); unit: kg] — The BW was evaluated after an overnight fast, through a bioimpedance digital scale results are reported in kilograms with a decimal.
  kg | 79.6 (11.9) | 79.1 (16.8) | 79.3 (14.3)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — The BMI was calculated by the square of the body height, and is universally expressed in units of kg/m2, resulting from mass in kilograms and height in metres.
  kg/m^2 | 31.1 (3.7) | 29.8 (5.2) | 30.4 (4.4)
Waist circumference (WC) [Mean (Standard Deviation); unit: cm] — The WC was evaluated after an overnight fast with a flexible tape in the midpoint between the lowest rib and the iliac crest and is expressed in centimeters.
  cm | 97.3 (6.9) | 98.8 (9.8) | 98 (8.3)
Systolic blood pressure (SBP) [Mean (Standard Deviation); unit: mmHg] — The SBP was evaluated with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures was considered as the value of SBP. The value was expressed on mmHg.
  mmHg | 117 (12) | 119 (12) | 118 (12)
Diastolic blood pressure (DBP) [Mean (Standard Deviation); unit: mmHg] — The DBP was evaluated with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures was considered as the value of DBP. The value was expressed on mmHg.
  mmHg | 77 (13) | 77 (8) | 77 (11)
Triglycerides (TGs) [Mean (Standard Deviation); unit: mmol/L] — The blood sample for determining of TGs, was taken after an overnight fast and was evaluated by spectrophotometry method. The value was expressed on mmol/L.
  mmol/L | 1.8 (1.3) | 1.5 (0.7) | 1.7 (1.0)
Total cholesterol (TC) [Mean (Standard Deviation); unit: mmol/L] — The blood sample for determining of TC, was taken after an overnight fast and was evaluated by spectrophotometry method. The value was expressed on mmol/L.
  mmol/L | 5.1 (0.1) | 5.2 (0.9) | 5.1 (0.9)
high-density lipoprotein cholesterol (HDL-C) [Mean (Standard Deviation); unit: mmol/L] | 1.0 (0.1) | 0.9 (0.3) | 0.9 (0.2)
Low-density lipoprotein cholesterol (LDL-C) [Mean (Standard Deviation); unit: mmol/L] — The blood sample for determining of LDL-C, was taken after an overnight fast and was calculated by Friedewald formula. The value was expressed on mmol/L.
  mmol/L | 3.5 (0.8) | 3.5 (0.5) | 3.5 (0.7)
Very-low density lipoprotein (VLDL) [Mean (Standard Deviation); unit: mmol/L] — The blood sample for determining the VLDL, was taken after an overnight fast and was calculated as triglycerides/5 . The value was expressed on mmol/L.
  mmol/L | 0.4 (0.3) | 0.3 (0.1) | 0.3 (0.2)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] — The blood sample for determining of FPG, was taken after an overnight fast and was evaluated by spectrophotometry method. The value was expressed on mmol/L.
  mmol/L | 5.9 (0.4) | 5.6 (0.4) | 5.8 (0.4)
2-hour postload plasma glucose (2-h PG) [Mean (Standard Deviation); unit: mmol/L] — The blood sample for determining of 2-h PG, was taken two hours after the ingestion of the drink with 75 g dextrose and was evaluated by spectrophotometry method. The value was expressed on mmol/L.
  mmol/L | 9.1 (1.2) | 8.6 (0.8) | 8.9 (1)
Glycated hemoglobin A1c [Mean (Standard Deviation); unit: Percent of glycated hemoglobin] | 5.8 (0.3) | 5.6 (0.2) | 5.7 (0.3)
Creatinine [Mean (Standard Deviation); unit: µmol/L] | 79.5 (17.7) | 70.8 (26.5) | 70.8 (17.7)
Area under the curve of glucose (AUCG) [Mean (Standard Deviation); unit: mmol/L/min] — The estimation for AUCG was calculated from parameters obtained during the 2 hours oral glucose tolerant test (OGTT) with 75 g dextrose by trapezoidal integration. The value was expressed mmol/L/min.
  mmol/L/min | 1157 (147) | 1078 (137) | 1120 (146)
Area under the curve of insulin (AUCI) [Mean (Standard Deviation); unit: pmol/L/min] — The estimation for AUCI was calculated from parameters obtained during the 2 hours oral glucose tolerant test (OGTT) with 75 g dextrose by trapezoidal integration. The value was expressed on pmol/L/min.
  pmol/L/min | 68,348 (20,329) | 63,544 (28,041) | 65946 (24188)
Total insulin secretion [Mean (Standard Deviation); unit: unitless] — Total insulin secretion was calculated with the insulinogenic index (ΔABC insulin / ΔABC glucose).
  unitless | 0.56 (0.20) | 0.54 (0.22) | 0.54 (0.22)
First phase of insulin secretion [Mean (Standard Deviation); unit: unitless] — First phase of insulin secretion was estimated using the Stumvoll index (1283+ 1.829 x insulin 30' - 138.7 x glucose 30' + 3.772 x insulin 0').
  unitless | 1297 (550) | 1391 (712) | 1344 (627)
Insulin sensitivity [Mean (Standard Deviation); unit: unitless] — Insulin sensitivity was calculated with Matsuda index [10,000 / √glucose 0' x insulin 0') (mean glucose oral glucose tolerance test (OGTT) x mean insulin OGTT)].
  unitless | 1.8 (0.8) | 2.5 (1.5) | 2.1 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Fasting Plasma Glucose
Description: After intervention by spectrophotometry
Time Frame: 90 days
Population: All participants, including those who dropped out before the end were taken into account for statical analysis (intention to treat).
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Gymnema Sylvestre | Placebo
Number analyzed (Participants) | 13 | 13
mmol/L | 77.4 (11.6) | 77.7 (13.2)

2. Primary Outcome: 2-hour Post Load Plasma Glucose (2-h PG)
Description: The blood sample for determining of 2-h PG, was taken two hours after the ingestion of the drink with 75 g dextrose and was evaluated by spectrophotometry method. The value was expressed on mmol/L.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Gymnema Sylvestre | Placebo
Number analyzed (Participants) | 13 | 13
mmol/L | 7.8 (1.7) | 7.9 (1.1)

3. Primary Outcome: Glycated Hemoglobin A1c (A1C)
Description: After intervention by high-performance liquid chromatography
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: Percent of glycated hemoglobin
Arm/Group | Gymnema Sylvestre | Placebo
Number analyzed (Participants) | 13 | 13
Percent of glycated hemoglobin | 5.4 (0.4) | 5.7 (0.5)

4. Primary Outcome: Total Insulin Secretion (Insulinogenic Index)
Description: Total insulin secretion was calculated with the insulinogenic index (ΔABC insulin / ΔABC glucose) after intervention.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Gymnema Sylvestre | Placebo
Number analyzed (Participants) | 13 | 13
Unitless | 0.51 (0.21) | 0.49 (0.18)

5. Primary Outcome: First Phase of Insulin Secretion
Description: First phase of insulin secretion was estimated using the Stumvoll index (1283+ 1.829 x insulin 30' - 138.7 x glucose 30' + 3.772 x insulin 0') after intervention.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Gymnema Sylvestre | Placebo
Number analyzed (Participants) | 13 | 13
Unitless | 1399 (552) | 1528 (677)

6. Primary Outcome: Insulin Sensitivity (Matsuda Index)
Description: Insulin sensitivity was calculated with Matsuda index [10,000 / √glucose 0' x insulin 0') (mean glucose oral glucose tolerance test (OGTT) x mean insulin OGTT)] after intervention.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Gymnema Sylvestre | Placebo
Number analyzed (Participants) | 13 | 13
Unitless | 2.4 (1.2) | 2.5 (1.2)

7. Secondary Outcome: Area Under the Curve of Glucose
Description: Area under the curve of glucose was obtained using the trapezoidal integration.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mmol/l/min
Arm/Group | Gymnema Sylvestre | Placebo
Number analyzed (Participants) | 13 | 13
mmol/l/min | 1075 (253) | 1018 (158)

8. Secondary Outcome: Area Under the Curve of Insulin
Description: After intervention area under the curve of insulin
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mmol/l/min
Arm/Group | Gymnema Sylvestre | Placebo
Number analyzed (Participants) | 13 | 13
mmol/l/min | 56968 (20787) | 53374 (20663)

9. Secondary Outcome: Body Weight (BW)
Description: The weight was measured at baseline, week 4, week 8 and week 12 with a bioimpedance balance and the entered values reflect the weight at week 12
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Gymnema Sylvestre | Placebo
Number analyzed (Participants) | 13 | 13
kg | 77.4 (11.6) | 77.7 (13.2)

10. Secondary Outcome: Body Mass Index (BMI)
Description: The Body Mass index was calculated at baseline and at week 12 with the Quetelet index and the entered values reflect the body mass index at week 12
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Gymnema Sylvestre | Placebo
Number analyzed (Participants) | 13 | 13
kg/m^2 | 30.3 (3.6) | 29.3 (4.4)

11. Secondary Outcome: Waist Circumference (WC)
Description: Waist circumference was evaluated at baseline and at week 12 with a flexible tape and the entered values reflects the waist circumference measure at week 12
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Gymnema Sylvestre | Placebo
Number analyzed (Participants) | 13 | 13
cm | 97.3 (7.7) | 99 (7.6)

12. Secondary Outcome: Systolic Blood Pressure (SBP)
Description: The Systolic Blood Pressure was evaluated at baseline and week 12 with a digital sphygmomanometer and the entered values reflect the blood pressure at week 12
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Gymnema Sylvestre | Placebo
Number analyzed (Participants) | 13 | 13
mmHg | 120 (15) | 120 (14)

13. Secondary Outcome: Diastolic Blood Pressure (DBP)
Description: The Diastolic blood pressure was evaluated at baseline and week 12 with a digital sphygmomanometer and the entered values reflect the blood pressure at week 12
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Gymnema Sylvestre | Placebo
Number analyzed (Participants) | 13 | 13
mmHg | 75 (10) | 77 (8)

14. Secondary Outcome: Total Cholesterol
Description: After intervention by spectrophotometry
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Gymnema Sylvestre | Placebo
Number analyzed (Participants) | 13 | 13
mmol/L | 4.7 (1.2) | 5.4 (1)

15. Secondary Outcome: Triglycerides
Description: After intervention by spectrophotometry
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Gymnema Sylvestre | Placebo
Number analyzed (Participants) | 13 | 13
mmol/L | 1.7 (0.9) | 1.6 (0.7)

16. Secondary Outcome: High Density Lipoprotein Cholesterol
Description: After intervention by spectrophotometry
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Gymnema Sylvestre | Placebo
Number analyzed (Participants) | 13 | 13
mmol/L | 0.9 (0.2) | 1.0 (0.3)

17. Secondary Outcome: Low Density Lipoprotein
Description: After intervention by spectrophotometry
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Gymnema Sylvestre | Placebo
Number analyzed (Participants) | 13 | 13
mmol/L | 2.5 (1.3) | 3.2 (1.6)

18. Secondary Outcome: Very Low Density Lipoprotein
Description: After intervention by spectrophotometry
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Gymnema Sylvestre | Placebo
Number analyzed (Participants) | 13 | 13
mmol/L | 0.3 (0.2) | 0.3 (0.1)

19. Secondary Outcome: Creatinine
Description: After intervention by spectrophotometry
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Gymnema Sylvestre | Placebo
Number analyzed (Participants) | 13 | 13
µmol/L | 70.8 (17.6) | 70.8 (17.6)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the 90 days of the study
Arm/Group | Gymnema Sylvestre | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 4/15 | 6/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gymnema Sylvestre (N=15) | Placebo (N=15)
Diarrea (Gastrointestinal disorders) | 4 | 2
Abdominal distention (Gastrointestinal disorders) | 4 | 6
Nausea (Gastrointestinal disorders) | 2 | 2
Anorexy (Gastrointestinal disorders) | 1 | 0
Sweet taste intolerance (Gastrointestinal disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 1
Polydipsia (General disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-01-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT02708966/Prot_SAP_ICF_000.pdf